CLINICAL TRIAL: NCT06989749
Title: Transcranial Direct Current Stimulation and Modulation of Affect and Pain
Acronym: StimMAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Responsible Party: Principal Investigator, Tor Wager, Diana L. Taylor Distinguished Professor, Trustees of Dartmouth College
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00032315
Record Dates: First submitted 2025-05-08; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: We Are Not Studying a Disease or Condition
Keywords: transcranial direct current stimulation; experimental pain; pain-related decision-making; social placebo effects
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Masking Description: Participants were blind to the tDCS type applied in each session. Personnel interacting directly with the study subjects are blind to the tDCS type in each session (Commonly known as "double blind"). Personnel analyzing data collected from the study are blind to the tDCS type applied in each session. Participants are blind to the exact temperatures (in Celsius) used in the study.
  Participants are blind to the temperatures received at the end of the decision making task.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Within-person Crossover (Other): This within-person crossover study involves a single arm, where each participant experiences an initial pain calibration session, followed by three full study sessions involving anodal, cathodal, or sham tDCS interventions. Only one intervention type (anodal, cathodal, or sham) is applied per session, in a randomized and double-blind fashion.
  Interventions: Other: Anodal tDCS; Other: Cathodal tDCS; Other: Sham tDCS

INTERVENTIONS:
Other: Anodal tDCS — Transcranial direct current stimulation (tDCS) is an experimental manipulation of brain circuitry using electrical current applied to the scalp. The equipment is commercially available (StarStim8, Neuroelectrics, Spain) and marketed for experimental research on brain function. Current is applied at 2 mA for 20 minutes. Electrodes are placed on the C3 and FP2 regions. There is a 30-second ramp-up and 30-second ramp-down of stimulation for each tDCS condition to minimize any discomfort during stimulation. In the anodal condition, real tDCS stimulation enters from the C3 electrode, and exits at the FP2 electrode.
  Other Names: Anodal Transcranial Direct Current Stimulation
Other: Cathodal tDCS — Transcranial direct current stimulation (tDCS) is an experimental manipulation of brain circuitry using electrical current applied to the scalp. The equipment is commercially available (StarStim8, Neuroelectrics, Spain) and marketed for experimental research on brain function. Current is applied at 2 mA for 20 minutes. Electrodes are placed on the C3 and FP2 regions. There is a 30-second ramp-up and 30-second ramp-down of stimulation for each tDCS condition to minimize any discomfort during stimulation. In the cathodal condition, real tDCS stimulation enters from the FP2 electrode, and exits at the C3 electrode.
  Other Names: Cathodal Transcranial Direct Current Stimulation
Other: Sham tDCS — This is the sham (or placebo) tDCS intervention. The tDCS device is applied for one minute, for a 30-second ramp-up and 30-second ramp-down of stimulation.
  Other Names: Sham Transcranial Direct Current Stimulation

SUMMARY:
This double-blind randomized crossover study aims to examine the effects of left primary motor cortex (M1) tDCS on evoked thermal pain perception, pain-related decision making, and placebo effects by manipulated pain and monetary offers accepted by others. The investigators plan to collect data for up to 50 participants who undergo four separate sessions: an initial pain calibration session and three experimental sessions with either anodal, cathodal, or sham tDCS. Each session includes pain testing before and after a single tDCS protocol (either anodal, cathodal, or sham), a pain-monetary decision-making task, and social placebo pain tests. All tasks following tDCS will take place inside the MR scanner. The investigators hypothesize that anodal M1 tDCS will decrease pain ratings, and that cathodal tDCS will increase them, both relative to the sham condition. The investigators will also examine the effects of M1 tDCS on social decision-making to examine whether it affects participants' valuation of pain and their altruistic behavior, as well as how these same factors impact pain sensation in the placebo task. The investigators hypothesize that participants will behave hyperaltruistically during the decision-making task, and that the same factors that influence choice will also impact pain perception in the same context.

DETAILED DESCRIPTION:
This study aims to examine the effects of M1 tDCS on induced experimental pain, pain-related decision making, and independently manipulate expectations based on the pain and monetary offered by others. This study involves 4 sessions, one thermal calibration session and three full study sessions where subjects will experience one of three tDCS conditions: anodal, cathodal, or sham. Participants receive only one condition of tDCS for each full session, and the order of which tDCS condition they receive is randomized. Participants are also asked to complete a decision-making task during each full study session, a Single-trial heat stimulation task based on the decision-making task, and finally a Social Decision Making and Placebo Responses task. Participants will complete all tasks following tDCS inside the MR scanner.

The initial pain calibration session is performed as a part of the screening process for each participant to ensure that all temperatures delivered during any subsequent procedures are within participants' tolerable range, and to obtain consent to participate in this research. The calibration procedure can improve the accuracy of the measurement because it adjusts the temperature based on the participants' reported sensation and allows for the determination of an individual's pain and tolerance level. Four runs (6 trials in each run and 24 trials totally) of noxious heat are administered to six forearm sites using iterative adaptive logistic regression. Each stimulus lasts 13 seconds, with 1.5 seconds for ramping. Sensation is rated on a circular scale from "no sensation" to "strongest imaginable". Participants report pain and tolerance with "yes" or "no" responses to "Painful?" and "Tolerate?" questions. The first calibration run familiarizes participants with 47°C heat on all sites. The second run includes 45°C, 47°C, and 48.9°C stimuli twice, randomly distributed. Runs three and four include low and high temperatures based on the pain and tolerance responses of previous trials. A logistic regression based on a 90% response to pain and tolerance of previous trials is used to determine the low and high threshold and is updated after each trial. After the final trial, low (pain) and high (tolerance) temperatures are determined using logistic regression across all trials, and three sites with the least mean absolute error values in rate-temperature linear regression are chosen for pain stimulation.

Each full session includes 3 run pains runs before tDCS, 20 min tDCS, 3 run pains tests after tDCS, Decision making task, and 3 runs of social decision making and placebo responses task. Each full session begins with three pain runs on three different regions of the right forearm (out of the 6 possible regions) used during the initial calibration session, and ends with three more pain runs on these same regions after tDCS. Each pain run consists of 12 trials using each participants' unique temperature range (pain and tolerance) obtained from the calibration session, such that there are 36 trials before tDCS, and 36 trials after tDCS.

The tDCS device is applied at 2 mA for 20 minutes using the StarStim system (Neuroelectrics, Spain). Electrodes are placed on the C3 and FP2 regions. There is a 30-second ramp-up and 30-second ramp-down of stimulation for each tDCS condition to minimize any discomfort during stimulation. During stimulation, a random fractal image is displayed on the participant's computer screen. Originally, the main purpose of presenting a random image during each tDCS stimulation was to facilitate a 1-month follow-up session for a memory test planned for future study. The assignment of pictures to task conditions is randomized for each participant and therefore picture identity is not confounded with task variables. After tDCS, participants complete a questionnaire related to sensations induced by tDCS.

Decision-making task During the initial phase of the decision-making task, participants are presented with 128 trials where they are given the option to either accept or reject offers for pain and monetary reward levels. The pain levels for the offers are randomized from 8 possible levels of each participant's own unique pain tolerance threshold (or 20%-90% of their tolerance), and the monetary rewards are also randomized from $1 to $8. The presentation order of the pain levels and monetary values for each offer are also randomized (e.g., $5 for 60%, or, 20% for $3, etc.). Participants are instructed that each monetary value represents 10 heat stimulation at that percentage of tolerance. The 128 offers are divided into two sets of 64 trials each, where the first set involves decisions about offers for oneself, while the second set involves decisions about offers for others. No heat stimulation is involved while participants complete the first phase of the task, and the trials are presented in blocks of 8 for each type. Upon completing the initial phase of the task, a random selection of trials decided for others are chosen, and the average reward value associated with the accepted trials among these trials is paid to the participants as compensation for their involvement in this task. In addition, one random trial from the decisions participants made for himself/herself is selected, and participants receive either 10 heat stimulation at that percent of tolerance and additional monetary value or no pain/monetary.

Social Decision Making and Placebo Responses Participants are also told during the second phase of this task that they will additionally receive three sets of 12 heat stimulation trials randomly selected from previous participants' decisions for future participants. Participants are first shown the decision from the previous participant (e.g., x. 50% tolerance paired with $4) and then receive a heat stimulation based on that offer. However, unbeknownst to participants, participants either receive a "high" or "low" temperature every trial in which the high temperature is always the participants maximum heat tolerance, and the low temperature is the maximum heat tolerance minus 1 degree celsius.

Full study sessions are scheduled with at least five days in between sessions, and roughly during the same time of day (e.g., morning, afternoon, evening, etc.).

ELIGIBILITY:
Inclusion Criteria:

* ages 18-55
* Participants must be capable of performing experimental tasks (e.g., are able to read)
* Fluent or native speakers of English

Exclusion Criteria:

* No self-reported current or history of depression, bipolar disorder, or other psychiatric diagnosis.
* No self-reported current seizure disorder (i.e., seizure within past 10 years)
* No history of stroke or other major neurological diagnosis.
* No self-reported current chronic pain, or acute pain within three months of the study period.
* No current migraine disorder (i.e., 15 headache days or more in 1 month).
* No use of central nervous system-effective medication or other medication for neurological/psychiatric treatment. No self-reported substance abuse within the last six months.
* No contraindication to MRI or tDCS (e.g., pregnancy, claustrophobia, pacemakers, ear/cochlear implants, shrapnel injuries, clips, or other ferromagnetic/electrical objects/devices, diagnosed brain abnormality such as tumor, or skin lesions on the scalp.).
* No contraindications for induced pain (e.g., no heart disease, high blood pressure, heart surgery, heart problems of any kind, severe asthma, respiratory problems of any kind, fibromyalgia, Raynaud's Syndrome or Disease, chronic pain, diabetes).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Pain Visual Analogue Scale | 3-10 sec post-stimulus throughout testing sessions, on average complete within 1 month
  Self-reported pain level following each thermal stimulus, measured on a visual analog scale. 0-100 scale with 0 indicating no pain and higher values indicating more pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth College, Hanover, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
Electronic data will be stored indefinitely and will not be shared with other investigators without explicit permission from the overseeing IRB.